CLINICAL TRIAL: NCT01849861
Title: Cardiopulmonary Capacity In Different Quartiles Ranges Of Reference For Serum Thyroid Stimulating Hormone (TSH): Sectional Evaluation And Effect Of The Use Of Methimazole In Elderly Population
Brief Title: Cardiopulmonary Capacity in Elderly With Different Ranges of Serum Thyroid Stimulating Hormone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Dhianah Santini de Oliveira Chachamovitz, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: idosos01
Record Dates: First submitted 2013-04-23; First posted 2013-05-09 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Cardiopulmonary Capacity; Ranges of TSH; Elderly Population
MeSH Terms: interventions — Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methimazole, (Experimental): Patients with serum TSH initially on the 1st. Quartile (TSH: 0.4 to 1.0 mIU / ml) will receive treatment with Methimazole (initial dose of 5mg/day) with the goal of raising the TSH values to range between 2.0 and 4.0 mIU / ml (the half upper range of normal).
  After six months with TSH in the target range (2.0 and 4.0 mIU / ml), these patients will be subjected to the same examination protocol performed at baseline and assessed to the effects of treatment on outcome variables.
  Variables considered in this study:
  * TSH and FT4
  * Questionnaire of Quality of life for older adults (WHOQOL-OLD)
  * Mini-Mental State Examination
  * Geriatric Depression Scale
  * Cardiopulmonary exercise testing - cardiopulmonary capacity
  Interventions: Drug: Methimazole

INTERVENTIONS:
Drug: Methimazole — Patients with serum TSH initially on the 1st. Quartile (TSH: 0.4 to 1.0 mIU / ml) will receive treatment with Methimazole (initial dose of 5mg/day) with the goal of raising the TSH values to range between 2.0 and 4.0 mIU / ml (the half upper range of normal).
  After six months with TSH in the target range (2.0 and 4.0 mIU / ml), these patients will be subjected to the same examination protocol performed at baseline and assessed to the effects of treatment on outcome variables.
  Variables considered in this study:
  * TSH and FT4
  * Questionnaire of Quality of life for older adults (WHOQOL-OLD)
  * Mini-Mental State Examination
  * Geriatric Depression Scale
  * Cardiopulmonary exercise testing - cardiopulmonary capacity
  Other Names: a single group

SUMMARY:
The purpose of this study is to correlate in an elderly population (≥ 65 years), the different levels of serum TSH, with cardiopulmonary capacity, quality of life, depressive symptoms and cognition. And assess whether the increased serum TSH to the upper half of the normal range, through the use of antithyroid drugs, is associated with improvements in these parameters.

DETAILED DESCRIPTION:
Specific Objectives:

Describe the cardiopulmonary capacity in elderly people with 65 years old or more, in different quartiles of normal range for serum TSH.

Assess the quality of life, mini mental health status and depression scale in seniors aged 65 or older, in different quartiles of normal range for serum TSH.

Quantify the possible effects related to the use of antithyroid drugs in cardiopulmonary capacity, quality of life, mini mental health status and depression scale in elderly people aged 65 or more, with the initial serum TSH at the lower limit of the normal range (1.0 milli-International unit/ml) (mIU/ml).

Justification:

Despite evidence that in the elderly population the mean serum TSH tends to be higher as compared to younger adults, there isn't a curve of normal range of TSH for this specific population (more shifted to the right, which would increase the number of diagnoses for subclinical hyperthyroidism).

Thus, elderly individuals, even when classified as euthyroidism, but presenting TSH in the normal lower range, may present at a greater risk of cardiovascular disease and therefore, may have indication for treatment.

These findings motivate and justify this study design, which may have great clinical relevance in the scientific community for its originality, and important clinical applicability.

Materials and Methods:

If the patient agrees to participate, an appointment will be scheduled at HUCFF that will be made: anamnesis, review of medical records, clinical examination and signing the Informed Consent Form (ICF).

Secondly, they will be guided and directed to: laboratory analysis for serum dosage of TSH and free thyroxine (FT4), cardiopulmonary exercise testing and application of the questionnaires of quality of life, mini mental health status and depression.

The study comprised of two parts:

Phase 1: Sectional:

* Analysis of variables.
* Sample as a whole and according to the quartiles of the reference range for serum TSH, with comparisons between groups.
* 1st Quartile: TSH: 0.4 to 1.0 mIU / ml.
* 2nd Quartile: TSH: 1.0 to 2.0 mIU / ml.
* 3rd Quartile: TSH: 2.0 to 3.0 mIU / ml.
* 4th Quartile: TSH: 3.0 to 4.0 mIU / ml Phase 2: Clinical uncontrolled. Patients with serum TSH initially on the 1st. Quartile (TSH: 0.4 to 1.0 mIU / ml) will receive treatment with Methimazole (initial dose of 5mg/day) with the goal of raising the TSH values to range between 2.0 and 4.0 mIU / ml (the half upper range of normal).

After six months with TSH in the target range (2.0 and 4.0 mIU / ml), these patients will be subjected to the same examination protocol performed at baseline and assessed to the effects of treatment on outcome variables.

Variables considered in this study:

* TSH and FT4
* Questionnaire of Quality of life for older adults (WHOQOL-OLD)
* Mini-Mental State Examination
* Geriatric Depression Scale
* Cardiopulmonary exercise testing - cardiopulmonary capacity Variables to be analyzed at rest, peak of the exercise and recovery: Heart rate, systolic blood pressure and diastolic blood pressure.

Variables to be assessed at peak effort: pulmonary ventilation, oxygen consumption, carbon dioxide production, ventilatory equivalent for oxygen and carbon dioxide, respiratory quotient, oxygen pulse, fraction of expired oxygen and carbon dioxide.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Healthy Men and women
* Registration at the University Hospital Clementino Fraga Filho (HUCFF).

Exclusion Criteria:

* Hypothalamic-pituitary disease
* Congestive cardiac insufficiency, chronic renal failure, acute renal failure, stroke, chronic obstructive pulmonary disease, asthma, cancer and / or cirrhosis.
* Diseases of the aorta, peripheral vascular disease, coronary artery disease (including angina, history of prior myocardial infarction or angina, or history of cardiac catheterization and angioplasty).
* Use of corticosteroids, amiodarone or dopamine, as well as any drug that interferes with the levels of thyroid hormones and / or thyroid function.
* Use of drugs that interfere with autonomic adaptation mechanism, such as beta-blockers, prolopa and calcium channel blockers. Hypertensive patients without use of such drugs may be included.
* Patients bedridden, wheelchair or with physical limitations (joint and muscle) to prevent the standing position for at least 20 minutes and the realization of the cardiopulmonary exercise test.
* Obesity with a body mass index equal or greater than 35 kg/m2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Correlate in a population of more than 65 years old, the different levels of serum TSH, with cardiopulmonary capacity and these effects from baseline after treatment with antithyroid drugs | six months
  Describe the cardiopulmonary capacity in elderly health population of 65 years old or more, in different quartiles of normal range for serum TSH.
  * Assess the outcome in the cardiopulmonary capacity in seniors aged 65 years old or more, in different quartiles of normal range for serum TSH.
  * Quantify the possible changes from baseline related to the use of antithyroid drugs in cardiopulmonary capacity in patients aged 65 or more, with the initial serum TSH at the lower limit of the normal range (1.0 mIU/ml)to values of TSH more than 2.0mUI/ml for six months.

SECONDARY OUTCOMES:
Assess the quality of life in seniors aged 65 years old or older, in different quartiles of normal range for serum TSH and these changes from baseline after use of methimazole | six months
  Describe the quality of life in elderly health population of 65 years old or more, in different quartiles of normal range for serum TSH.
  * Assess the outcome in quality of life in seniors aged 65 olde or more, in different quartiles of normal range for serum TSH
  * Quantify the possible changes from baseline related to the use of antithyroid drugs in quality of life in patients aged 65 or more, with the initial serum TSH at the lower limit of the normal range (1.0 mIU/ml)to values of TSH more than 2.0mUI/ml for six months..
Assess the mini mental health status in seniors aged 65 years old or older, in different quartiles of normal range for serum TSH and these changes from baseline after use of methimazole | six months
  Describe the mini mental health status in elderly health population of 65 years old or more, in different quartiles of normal range for serum TSH.
  * Assess the outcome in mini mental health status in seniors aged 65 olde or more, in different quartiles of normal range for serum TSH.
  * Quantify the possible changes from baseline related to the use of antithyroid drugs in mini mental health status in patients aged 65 or more, with the initial serum TSH at the lower limit of the normal range (1.0 mIU/ml)to values of TSH more than 2.0mUI/ml for six months.
Assess the depression scale in seniors aged 65 years old or older, in different quartiles of normal range for serum TSH and these changes from baseline after use of methimazole | six months
  Describe the depression scale in elderly health population of 65 years old or more, in different quartiles of normal range for serum TSH.
  * Assess the outcome in depression scale in seniors aged 65 olde or more, in different quartiles of normal range for serum TSH.
  * Quantify the possible changes from baseline related to the use of antithyroid drugs in the depression scale in patients aged 65 years old or more, with the initial serum TSH at the lower limit of the normal range (1.0 mIU/ml)to values of TSH more than 2.0mUI/ml for six months..

CONTACTS AND LOCATIONS:
Overall Officials: Dhiãnah SO Chachamovitz, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil